CLINICAL TRIAL: NCT02807506
Title: PFI: BIC Affordable and Mobile Assistive Robots for Elderly Care
Brief Title: Affordable Mobile Robots for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 820915
Record Dates: First submitted 2016-03-31; First posted 2016-06-21 (Estimated); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Aging
Keywords: elders; robotics; low income population; activities of daily living; instrumental activities of daily living; social robotics; stroke; aged; Retirement; Housing for elderly; Homes for the aged
MeSH Terms: conditions — Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Aim 1 (Survey): Elders (Experimental): Observe Elders, Clinicians and Caregiver's survey, interview and observational responses to stage-wise experimental deployments of a mobile service robot - 1st concept (elders, clinicians, caregivers), 2nd mobile base (elders only), and 3rd mobile base with arm in daily supportive tasks (elders only)
  Interventions: Other: Survey
- Aim 1 (Survey): Clinicians (Experimental): Observe Elders, Clinicians and Caregiver's survey, interview and observational responses to stage-wise experimental deployments of a mobile service robot - 1st concept (elders, clinicians, caregivers), 2nd mobile base (elders only), and 3rd mobile base with arm in daily supportive tasks (elders only)
  Interventions: Other: Survey
- Aim 1 (Survey): Caregivers (Experimental): Observe Elders, Clinicians and Caregiver's survey, interview and observational responses to stage-wise experimental deployments of a mobile service robot - 1st concept (elders, clinicians, caregivers), 2nd mobile base (elders only), and 3rd mobile base with arm in daily supportive tasks (elders only)
  Interventions: Other: Survey
- Aim 2: Deployment 1 (Elders) (Experimental): Observe Elders, Clinicians and Caregiver's survey, interview and observational responses to stage-wise experimental deployments of a mobile service robot - 1st concept (elders, clinicians, caregivers), 2nd mobile base (elders only), and 3rd mobile base with arm in daily supportive tasks (elders only)
  Interventions: Device: Mobile Service Robot
- Aim 2: Deployment 2 (Elders) (Experimental): Observe Elders, Clinicians and Caregiver's survey, interview and observational responses to stage-wise experimental deployments of a mobile service robot - 1st concept (elders, clinicians, caregivers), 2nd mobile base (elders only), and 3rd mobile base with arm in daily supportive tasks (elders only)
  Interventions: Device: Mobile Service Robot

INTERVENTIONS:
Device: Mobile Service Robot — The goal is to build a low-cost mobile service robot with an arm that will focus on the simple, but key, repetitive, data-driven tasks that robots do well. Rather than attempt to create a robot helper that mimics humans, the goal is to free human caregivers from the time-consuming tasks that robots can accomplish with facility, thereby allowing humans to focus on tasks that humans do best (i.e. human contact).
  Arms: Aim 2: Deployment 1 (Elders); Aim 2: Deployment 2 (Elders)
Other: Survey — Observe Elders, Clinicians and Caregiver's survey, interview and observational responses to stage-wise experimental deployments of a mobile service robot.
  Arms: Aim 1 (Survey): Caregivers; Aim 1 (Survey): Clinicians; Aim 1 (Survey): Elders

SUMMARY:
This project develops and tests the use of service robots to track health of the elderly over time. The objectives are to develop a low-cost mobile manipulator capable of a limited set of elder- relevant manipulation tasks (e.g. picking up dropped items). The investigators will visualize and model the use of the service robot during deployments at an elder care facility. Feedback from focus groups with elders and clinicians will inform the necessary engineering innovation.

DETAILED DESCRIPTION:
The goal is to develop in three stages a new affordable robot with the participation of Living Independently for Elders (LIFE) members and clinicians. The robot will be developed by a multidisciplinary team headed by Dr. Yim at University of Pennsylvania (UPENN) (PI), Dr. Tessa Lau at Savioke Corp, and Drs. Johnson and Cacchionne at UPENN PM&R and UPENN Nursing, respectively. The aim is to build a low-cost robot platform that will focus on the simple, but key, repetitive, data-driven tasks that robots do well. Rather than attempt to create a robot helper that mimics humans, the aim is to free human caregivers from the time-consuming tasks that robots can accomplish with facility, thereby allowing humans to focus on tasks that humans do best (i.e. human contact). Participatory reviews of the developed prototypes will be completed at each stage (each year) with the LIFE members and clinicians. There are three research questions the investigators hope to answer all while building an effective system to synergistically satisfy the business needs:

R1) Although activities of daily living (ADLs) for elder health have previously been documented and categorized, no research has been done to characterize them from the perspective of their feasibility of automation using an affordable mobile manipulation robot. How can known ADLs be characterized according to how much they would benefit from robotic assistance given varying levels of robot capabilities (mobility, limited manipulation, full manipulation)?

R2) A manipulator arm must be safe, affordable, and performant enough to assist in ADLs for elder heath. What new breakthroughs are required to develop new manipulation technology that satisfies these constraints?

R3) A data-driven service robotics What are the concomitant key usability and acceptance of service features required system has the potential to affect elder health in a positive way. How can predictive service robotics best be used to maintain and improve elder health? Which specific robot behaviors have the most impact on elders' well-being?

ELIGIBILITY:
Inclusion Criteria:

* Elders, age 55 and older,who are members of Living Independently For Elders (LIFE) run by the University of Pennsylvania, School of Nursing and their caregivers.
* Elders at Kearsley or Mercy Douglas who are 62 years and older, in imminent risk of a nursing home placement, attends LIFE center daily (day program), able to have activities of daily living (ADL) needs met by caregivers, able to pay required rent for apartment, and able to function safely in community with other elders.
* Savioke may conduct additional focus groups at The Forum at Rancho San Antonio a Continuing Care Retirement Community located in Silicon Valley.
* Clinicians will be recruited from the clinical staff working at LIFE, Kearsley, and Mercy Douglas which consists of primary care physicians, nurses and nurse practitioners, licensed social workers, and physical and occupational therapists.
* Caregivers will be recruited from the clinical staff working at LIFE, Kearsley, and Mercy Douglas which consists of certified nursing assistants (CNAs).

Exclusion Criteria:

* Unable to cognitively give consent
* Unable to understand the study or refuse to comply with procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-07; Primary Completion 2021-06-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Johnson, PhD, Principal Investigator — University of Pennsylvania; Mark Yim, PhD, Principal Investigator — University of Pennsylvanica
Locations (1):
- Mercy Living Independently for Elders (L.I.F.E) - West Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mucchiani C, Torres WO, Edgar D, Johnson MJ, Cacchione PZ, Yim M. Development and deployment of a mobile manipulator for assisting and entertaining elders living in supportive apartment living facilities. In2018 27th IEEE International Symposium on Robot and Human Interactive Communication (RO-MAN) 2018 Aug 27 (pp. 121-128). IEEE.
- [Background] Mucchiani C, Cacchione P, Johnson M, Mead R, Yim M. Deployment of a Socially Assistive Robot for Assessment of COVID-19 Symptoms and Exposure at an Elder Care Setting. In2021 30th IEEE International Conference on Robot & Human Interactive Communication (RO-MAN) 2021 Aug 8 (pp. 1189-1195). IEEE.
- [Background] Cacchione, P., Mucchiani, C., Lima, K., Mead, R., Yim, M. and Johnson, M., 2020. Engaging End Users in Designing Systems and Hardware for a Socially Assistive Robot. Innovation in Aging, 4(Suppl 1), pp.823-823.
- [Result] Johnson MJ, Johnson MA, Sefcik JS, Cacchione PZ, Mucchiani C, Lau T, Yim M. Task and design requirements for an affordable mobile service robot for elder care in an all-inclusive care for elders assisted-living setting. International journal of social robotics. 2020 Nov;12(5):989-1008.
- [Result] Mucchiani C, Sharma S, Johnson M, Sefcik J, Vivio N, Huang J, Cacchione P, Johnson M, Rai R, Canoso A, Lau T. Evaluating older adults' interaction with a mobile assistive robot. In2017 IEEE/RSJ International Conference on Intelligent Robots and Systems (IROS) 2017 Sep 24 (pp. 840-847). IEEE.
- [Result] Sefcik JS, Johnson MJ, Yim M, Lau T, Vivio N, Mucchiani C, Cacchione PZ. Stakeholders' Perceptions Sought to Inform the Development of a Low-Cost Mobile Robot for Older Adults: A Qualitative Descriptive Study. Clin Nurs Res. 2018 Feb;27(1):61-80. doi: 10.1177/1054773817730517. Epub 2017 Sep 16. PMID 28918654
- [Result] Mucchiani C, Cacchione P, Torres W, Johnson MJ, Yim M. Exploring low-cost mobile manipulation for elder care within a community based setting. Journal of Intelligent & Robotic Systems. 2020 Apr;98(1):59-70.
- See also: Article about robot for eldercare — http://www.nsf.gov/discoveries/disc_summ.jsp?cntn_id=138849

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Elders, caregivers, and clinicians were recommended and recruited to the study from the same recruitment site.
Groups:
- Aim 1 (Survey): Elders; Aim 1 (Survey): Clinicians; Aim 1 (Survey): Caregivers: Observe Elders, Clinicians and Caregiver's survey, interview and observational responses to stage-wise experimental deployments of a mobile service robot.
- Aim 2: Deployment 1 (Elders); Aim 2: Deployment 2 (Elders): Observe Elders responses to stage-wise experimental deployments of a mobile service robot - 1st concept (elders, clinicians, caregivers), 2nd mobile base (elders only), and 3rd mobile base with arm in daily supportive tasks (elders only)
Period: Aim 1: Survey
Arm/Group | Aim 1 (Survey): Elders | Aim 1 (Survey): Clinicians | Aim 1 (Survey): Caregivers | Aim 2: Deployment 1 (Elders) | Aim 2: Deployment 2 (Elders)
Started | 5 | 8 | 6 | 0 | 0
Completed | 5 | 8 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Aim 2: Deployment 1
Arm/Group | Aim 1 (Survey): Elders | Aim 1 (Survey): Clinicians | Aim 1 (Survey): Caregivers | Aim 2: Deployment 1 (Elders) | Aim 2: Deployment 2 (Elders)
Started | 0 | 0 | 0 | 16 | 0
Completed | 0 | 0 | 0 | 16 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Aim 2: Deployment 2
Arm/Group | Aim 1 (Survey): Elders | Aim 1 (Survey): Clinicians | Aim 1 (Survey): Caregivers | Aim 2: Deployment 1 (Elders) | Aim 2: Deployment 2 (Elders)
Started | 0 | 0 | 0 | 0 | 18
Completed | 0 | 0 | 0 | 0 | 18
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 39 elders, 8 clinicians, 6 caregivers
Groups:
- Clinicians, Caregivers and Elders: Observe Elders, Clinicians and Caregiver's survey, interview and observational responses to stage-wise experimental deployments of a mobile service robot - 1st concept, 2nd mobile base, and 3rd mobile base with arm in daily supportive tasks
  Mobile Service Robot: The goal is to build a low-cost mobile service robot with an arm that will focus on the simple, but key, repetitive, data-driven tasks that robots do well. Rather than attempt to create a robot helper that mimics humans, the goal is to free human caregivers from the time-consuming tasks that robots can accomplish with facility, thereby allowing humans to focus on tasks that humans do best (i.e. human contact).
Arm/Group | Clinicians, Caregivers and Elders
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants] — Population: Each demographic group that was analyzed in the Arm group
  Participants
    Elders: number analyzed (Participants) | 39
    Elders: <=18 years | 0
    Elders: Between 18 and 65 years | 6
    Elders: >=65 years | 33
    Clinicians: number analyzed (Participants) | 8
    Clinicians: <=18 years | 0
    Clinicians: Between 18 and 65 years | 8
    Clinicians: >=65 years | 0
    Caregivers: number analyzed (Participants) | 6
    Caregivers: <=18 years | 0
    Caregivers: Between 18 and 65 years | 6
    Caregivers: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Each demographic group that was analyzed in the Arm group
  Participants
    Elders: number analyzed (Participants) | 39
    Elders: Female | 21
    Elders: Male | 18
    Clinicians: number analyzed (Participants) | 8
    Clinicians: Female | 7
    Clinicians: Male | 1
    Caregivers: number analyzed (Participants) | 6
    Caregivers: Female | 6
    Caregivers: Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each demographic group that was analyzed in the Arm group
  Participants
    Elders: number analyzed (Participants) | 39
    Elders: American Indian or Alaska Native | 0
    Elders: Asian | 0
    Elders: Native Hawaiian or Other Pacific Islander | 0
    Elders: Black or African American | 38
    Elders: White | 0
    Elders: More than one race | 0
    Elders: Unknown or Not Reported | 1
    Clinicians: number analyzed (Participants) | 8
    Clinicians: American Indian or Alaska Native | 0
    Clinicians: Asian | 0
    Clinicians: Native Hawaiian or Other Pacific Islander | 0
    Clinicians: Black or African American | 1
    Clinicians: White | 7
    Clinicians: More than one race | 0
    Clinicians: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 6
    Caregivers: American Indian or Alaska Native | 0
    Caregivers: Asian | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0
    Caregivers: Black or African American | 6
    Caregivers: White | 0
    Caregivers: More than one race | 0
    Caregivers: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Usability Scale for Deployment 1
Description: Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) assistance, feasibility of automation of manipulator and arm measured by surveys and observation of participants in focus group. Usability of robot system for walking and water delivery tasks. Usability survey scored from 0 to 100, with 100 being the most favorable response. A number greater than 68 is good.
Time Frame: 1 session, about 1 hour in length
Population: Elders above the age of 55 years old who participated in the water delivery and walking tasks (Aim 2, Deployment 1).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aim 2: Deployment 1 (Elders): Water delivery and walking tasks
Arm/Group | Aim 2: Deployment 1 (Elders)
Number analyzed (Participants) | 16
score on a scale
  Water Delivery with Robot: number analyzed (Participants) | 8
  Water Delivery with Robot | 78.13 (3.608)
  Walking Delivery Task with Robot: number analyzed (Participants) | 12
  Walking Delivery Task with Robot | 77.08 (4.167)

2. Primary Outcome: Usability Scale for Deployment 2
Description: Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) assistance, feasibility of automation of manipulator and arm measured by surveys and observation of participants in focus group. Usability of robot system for walking and water delivery tasks. Usability survey scored out of 7. Users ranked tasks on a scale of 1-7, 7 being very usable.
Time Frame: 1 session, about 1 hour in length
Population: Elders above the age of 55 years old who participated in the gaming tasks (Aim 2, Deployment 2).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aim 2: Deployment 2 (Elders): Gaming Task
Arm/Group | Aim 2: Deployment 2 (Elders)
Number analyzed (Participants) | 18
score on a scale | 6.266 (1.204)

3. Primary Outcome: Sociability Scale for Deployment 1
Description: Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) assistance, feasibility of automation of manipulator and arm measured by surveys and observation of participants in focus group. Sociability of robot system for walking and water delivery tasks. Sociability survey scored from 0 to 100, with 100 being the most favorable response. A number greater than 68 is good.
Time Frame: 1 session, about 1 hour in length
Population: Elders above the age of 55 years old who participated in the water delivery and walking tasks (Aim 2, Deployment 1).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 2: Deployment 1 (Elders)
Number analyzed (Participants) | 16
score on a scale
  Water Delivery Task with Robot: number analyzed (Participants) | 8
  Water Delivery Task with Robot | 59.38 (11.97)
  Walking Task with Robot: number analyzed (Participants) | 12
  Walking Task with Robot | 82.29 (10.96)

4. Primary Outcome: Sociability Scale for Deployment 2
Description: Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) assistance, feasibility of automation of manipulator and arm measured by surveys and observation of participants in focus group. Sociability of robot system for walking and water delivery tasks. Sociability survey scored out of 7. Users ranked tasks on a scale of 1-7, 7 being very usable.
Time Frame: 1 session, about 1 hour in length
Population: Elders above the age of 55 years old who participated in the gaming tasks (Aim 2, Deployment 2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 2: Deployment 2 (Elders)
Number analyzed (Participants) | 18
score on a scale | 6.882 (0.332)

5. Primary Outcome: Acceptability Scale for Deployment 1
Description: Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) assistance, feasibility of automation of manipulator and arm measured by surveys and observation of participants in focus group. Acceptability of robot system for walking and water delivery tasks. Acceptability survey scored from 0 to 100, with 100 being the most favorable response. A number greater than 68 is good.
Time Frame: 1 session, about 1 hour in length
Population: Elders above the age of 55 years old who participated in the water delivery and walking tasks (Aim 2, Deployment 1).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 2: Deployment 1 (Elders)
Number analyzed (Participants) | 16
score on a scale
  Water Delivery Task with Robot: number analyzed (Participants) | 8
  Water Delivery Task with Robot | 76.56 (15.63)
  Walking Task with Robot: number analyzed (Participants) | 12
  Walking Task with Robot | 82.29 (7.116)

6. Primary Outcome: Acceptability Scale for Deployment 2
Description: Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) assistance, feasibility of automation of manipulator and arm measured by surveys and observation of participants in focus group. Acceptability of robot system for walking and water delivery tasks. Acceptability survey scored out of 7. Users ranked tasks on a scale of 1-7, 7 being very usable.
Time Frame: 1 session, about 1 hour in length
Population: Elders above the age of 55 years old who participated in the gaming tasks (Aim 2, Deployment 2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 2: Deployment 2 (Elders)
Number analyzed (Participants) | 18
score on a scale | 6.608 (1.056)

ADVERSE EVENTS:
Time Frame: Approximately 1 hour (duration of participation session)
Arm/Group | Clinicians, Caregivers and Elders
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT02807506/Prot_000.pdf
  • Informed Consent Form (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT02807506/ICF_001.pdf